CLINICAL TRIAL: NCT02490202
Title: A Randomized, Placebo-controlled, Prospective, Double-blind, Multicenter Phase 2/3 Study of the Efficacy and Safety of SANGUINATE™ for Reduction of Delayed Graft Function in Recipients of a Donation After Brain Death Kidney Transplant
Brief Title: Efficacy and Safety of SANGUINATE™ for Reduction of Delayed Graft Function in Patients Receiving a Kidney Transplant
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGTP-002
Record Dates: First submitted 2015-06-16; First posted 2015-07-03 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Delayed Function of Renal Transplant
MeSH Terms: interventions — PEGylated carboxyhemoglobin bovine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SANGUINATE (Experimental): Two (2) infusions of SANGUINATE
  Interventions: Drug: SANGUINATE
- Normal Saline (Placebo Comparator): Two (2) infusions of Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: SANGUINATE — Two (2) infusions of 320 mg/kg of SANGUINATE at Baseline and Day 1
  Other Names: pegylated carboxyhemoglobin bovine
  Arms: SANGUINATE
Drug: Normal Saline — Two (2) infusions of Normal Saline at an equal volume to SANGUINATE at Baseline and Day 1.
  Arms: Normal Saline

SUMMARY:
Safety and efficacy study of SANGUINATE on reduction of delayed graft function (DGF) in patients who will be recipients of a donation after brain death (DBD) donor kidney.

DETAILED DESCRIPTION:
Phase 2: Sixty (60) adult subjects who will be recipients of a donation after brain death (DBD) donor kidney and who meet all eligibility criteria will be randomized 1:1 within 48 hours prior to transplant surgery to receive: two infusions of SANGUINATE at a dose of 320 mg/kg or placebo on the day of surgery and approximately 24 hours after surgery. Patients will be hospitalized for up to 5 days and the study duration will be 30 days. Results will be used to inform the study design characteristics for Phase III, including sample size.

Phase III: The same inclusion/exclusion requirements, dosing schedule, hospitalization stay and outpatient visits as in Phase II with additional visits scheduled at Day 90, Day 180 and Day 365. Study duration will be 365 days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide written informed consent.
2. Male or female subject at least 18 years of age.
3. Dialysis-dependent renal failure initiated at least 3 months prior to transplantation.
4. Subject is to be the recipient of a first kidney transplant from a deceased donor (brain death criteria).
5. Is able to receive intravenous infusions of study drug.
6. Anticipated donor organ cold ischemia time < 30 hours.
7. A calculated prediction of DGF risk of least 25%.
8. Females of childbearing potential must agree to use 2 forms of effective birth control regimen (at least one-barrier method) during the initial 30-day study period.
9. Male subjects must agree to use condoms or other suitable means of pregnancy prevention.

Exclusion Criteria:

1. Has received a blood transfusion of packed red blood cells (PRBC), other than with leukocyte-poor blood, within the 90-day period prior to screening.
2. Recipient of a live donor kidney or a kidney from a donation after cardiac death (DCD) donor.
3. Recipient of donor kidney preserved with normothermic machine perfusion.
4. Is scheduled to undergo multi-organ transplantation.
5. Has planned transplant of kidney(s) from a donor < 6 years of age.
6. Has planned transplant of kidneys that are implanted en bloc (dual kidney transplant).
7. Has planned transplant of dual kidneys (from the same donor) transplanted not en bloc.
8. Body Mass Index (BMI) > 38 kg/m2
9. Is scheduled for transplantation of a kidney from a donor who is known to have received an investigational therapy (under another Investigational New Drug) for ischemic/reperfusion injury immediately prior to organ recovery.
10. Is scheduled to receive an blood type-incompatible donor kidney.
11. Has undergone desensitization to remove antibodies prior to transplantation.
12. Total bilirubin > 1.5 mg per dL, transaminase more than twice the upper limit of normal or evidence of hepatic insufficiency
13. Has participated in an investigational study within the last 30 days or received an investigational product within 5 half-lives of the study drug administration, whichever is longest. Potential subjects participating in a strictly observational study or a study involving approved treatments should be discussed with the Medical Monitor.
14. Has a history of human immunodeficiency virus (HIV)
15. History or presence of active substance abuse (illicit drugs or alcohol) in the previous 6 months, as believed by the Investigator
16. Presence of ECG-based evidence of acute myocardial infarction, unstable angina, decompensated heart failure, third degree heart block or cardiac arrhythmia associated with hemodynamic instability
17. History or presence of any disease or psychiatric condition that in the Investigator's assessment that would increase the risk to subjects associated with study participation, drug administration or interpretation of results
18. History of biopsy-confirmed malignancy within 5 years of randomization, with the exception of adequately treated basal cell or squamous cell carcinoma in situ skin lesions, carcinoma of the cervix in situ, or early detected prostate cancer.
19. Female subject who is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction of delayed graft function (DGF) | 30 Days
  Reduction of delayed draft function will be measured by the number of dialysis sessions.
Participants With at Least One Occurrence of Safety Composite Endpoint by Treatment Group | Phase 2 - 30 Days; Phase 3: Safety - 90 days; Serious Adverse Events and Adverse Events of Special Interest - 180 Days; Graft Survival - 365 Days
  Composite endpoint defined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis, graft loss, death and other reported adverse events

SECONDARY OUTCOMES:
Proportion of subjects requiring dialysis for any reason in the first 7 days post-transplant | 7 Days
Proportion of subjects requiring dialysis only in the first 5 days post-transplant | 5 Days
Number of days of dialysis therapy. | 30 Days
Proportion of subjects with a fall in serum creatinine. | 7 Days
Proportion of subjects with a serum creatinine greater than 3 mg/dL, but who did not require dialysis by Day 5 post-transplant | 5 Days
Rate of change in estimated creatinine clearance and estimated glomerular filtration rate over time | Phase 2: 30 Days

OTHER OUTCOMES:
Determination of sample size for Phase 3 based upon the results from Phase 2. | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Misra, PhD, Study Director — Prolong Pharmaceuticals
Locations (20):
- United States (20):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - California Institute of Renal Research, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Medstar Georgetown University Hosiptal, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - UIC University of Illinois at Chicago, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - Central Pennsylvania Transplant Foundation, Harrisburg, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No